CLINICAL TRIAL: NCT05842538
Title: Robotic Assisted Surgery In Total Knee Replacement Versus Manual Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Robotic Assisted Surgery In Total Knee Replacement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Principal Investigator, Maziar Mohaddes Ardebili, Associate Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAKER
Record Dates: First submitted 2022-10-03; First posted 2023-05-06 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAKO TKA (Experimental)
  Interventions: Device: Triathlon
- Conventional (Active Comparator)
  Interventions: Device: Triathlon

INTERVENTIONS:
Device: Triathlon — Total knee arthroplasty

SUMMARY:
The goal of this clinical trial is to compare robotic arm assisted surgery with manual surgery in patients operated with knee replacement.

The main aim of the study is to compare changes in joint awareness (measured by the Forgotten Joint Score.

Participants who are listed for knee arthroplasty are randomised to either robotic arm assisted surgery or manual surgery.

DETAILED DESCRIPTION:
Study Title:

Robotic Assisted Surgery in total knee replacement versus Manual Total Knee Arthroplasty: A randomised controlled trial

Type of study:

CE marked device study

Trial Design:

Multi-center site prospective parallel group randomised controlled trial

Trial Participants:

Listed for routine primary total knee replacements

Investigational Device:

MAKO Robotic Arm Assisted Surgical System

Control:

Conventional jig-based surgery

Implant (Intervention and Control):

Triathlon TKR

Planned Sample Size:

200 (100 MAKO, 100 Manual)

Follow-up duration:

24 months following surgery

Planned Trial Period:

Nov 2022 - 2024

Primary Objective:

To compare changes in joint awareness (measured by the Forgotten Joint Score (FJS)20) from baseline to 12 months following TKR between the two groups.

Secondary Objectives

1. To compare pain measured using the pain visual analogue scale.
2. To compare the health-related quality of life using the EQ5D-3L at baseline, 3, 12 and 24 months.
3. To compare changes in knee function in activities of daily living (measured by the Oxford knee score (OKS)19) from baseline to 3, 12 and 24 months.
4. To compare changes in clinically assessed pain and stiffness (measured by the Knee Society Score (KSS)) at baseline to 3 and 12 months.
5. To compare revision rate using implant migration measured by CTMA at 12 and 24 months as a surrogate marker for revision.

Primary Endpoint:

Functional outcome measured by the changes in joint awareness of the FJS score at 12 months following the intervention.

Secondary Endpoints:

Secondary outcomes will be collected up to 24 months following the intervention.

Device Name:

Both arms will receive Triathlon TKR with a highly crossed linked (X3) cruciate retaining polyethylene insert.

The intervention group will utilise the MAKO robotic arm to make the bone cuts.

ELIGIBILITY:
Inclusion Criteria:

* Listed for elective primary TKR for end stage osteoarthritis
* Suitable candidate for a cruciate retaining TKR (Triathlon prosthesis)
* Male or Female, aged 18 years or above (18-80 at the time of listing for surgery).
* Able to understand and provide written consent.

Exclusion Criteria:

* Varus deformity of > 20 degrees observed by consultant on examination
* Patient is unable to comply with the study protocol (incl. refusal for CT scan)
* Female participant who is pregnant, lactating or planning pregnancy during the course of the study.
* Requires patella resurfacing
* Inability to understand the patient information for the study, provide written informed consent or answer study questionnaires for cognitive or language reasons
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Forgotten Joint Score | 1 year
  Patient-reported outcome

SECONDARY OUTCOMES:
Knee pain | 2 years
  Patient-reported outcome
EQ-5D | 3, 12, 24 months
  Patient-reported outcome
Oxford Knee Score | 3, 12, 24 months
  Patient-reported outcome
Knee Society Score | 3, 12, 24 months
  Physician-reported outcome

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Sahlgrenska University hospital, Gothenburg
  - Örebro University Hospital, Department of Medical Sciences, Örebro

IPD SHARING:
Plan to Share IPD: No